CLINICAL TRIAL: NCT03162783
Title: A Single-Center, Phase 2a, Randomized, Double Masked, Clinical Study to Assess the Safety, Tolerability, and Pharmacodynamic Activity of ADX-102 Ophthalmic Solution in Subjects With Dry Eye Syndrome
Brief Title: A Randomized, Double Masked, Clinical Study of Subjects With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ADX-102-DES-007
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2018-06

CONDITIONS: Dry Eye Syndromes
Keywords: Aldeyra
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADX-102 Ophthalmic Solution (0.5%) (Experimental)
  Interventions: Drug: ADX-102 Ophthalmic Solution (0.5%)
- ADX-102 Ophthalmic Solution (0.1%) (Experimental)
  Interventions: Drug: ADX-102 Ophthalmic Solution (0.1%)
- ADX-102 Ophthalmic Lipid Solution (0.5%) (Experimental)
  Interventions: Drug: ADX-102 Ophthalmic Lipid Solution (0.5%)

INTERVENTIONS:
Drug: ADX-102 Ophthalmic Solution (0.5%) — ADX-102 Ophthalmic Solution (0.5%) administered for approximately 4 weeks.
  Arms: ADX-102 Ophthalmic Solution (0.5%)
Drug: ADX-102 Ophthalmic Solution (0.1%) — ADX-102 Ophthalmic Solution (0.1%) administered for approximately 4 weeks.
  Arms: ADX-102 Ophthalmic Solution (0.1%)
Drug: ADX-102 Ophthalmic Lipid Solution (0.5%) — ADX-102 Ophthalmic Lipid Solution administered for approximately 4 weeks.
  Arms: ADX-102 Ophthalmic Lipid Solution (0.5%)

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and pharmacodynamic activity of ADX-102 Ophthalmic Solutions and ADX-102 Ophthalmic Lipid Solution in subjects with dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age of either gender and any race;
* Have a reported history of dry eye for at least 6 months prior to Visit 1;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used cyclosporine 0.05% or lifitegrast 5.0% ophthalmic solution within 45 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within the last 6 months;
* Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clark D, Sheppard J, Brady TC. A Randomized Double-Masked Phase 2a Trial to Evaluate Activity and Safety of Topical Ocular Reproxalap, a Novel RASP Inhibitor, in Dry Eye Disease. J Ocul Pharmacol Ther. 2021 May;37(4):193-199. doi: 10.1089/jop.2020.0087. Epub 2021 Jan 15. PMID 33450164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | ADX-102 Ophthalmic Solution (0.1%) | ADX-102 Ophthalmic Lipid Solution (0.5%)
Started | 17 | 17 | 17
Completed | 12 | 16 | 11
Not Completed | 5 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | ADX-102 Ophthalmic Solution (0.1%) | ADX-102 Ophthalmic Lipid Solution (0.5%) | Total
Number analyzed (Participants) | 17 | 17 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 4 | 18
  >=65 years | 10 | 10 | 13 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 11 | 34
  Male | 3 | 8 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 15 | 17 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 16 | 15 | 17 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Iris Color (Right Eye) [Number; unit: participants]
  Black | 0 | 0 | 0 | 0
  Blue | 7 | 2 | 5 | 14
  Brown | 6 | 13 | 6 | 25
  Hazel | 3 | 1 | 4 | 8
  Green | 1 | 1 | 2 | 4
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Number; unit: participants]
  Black | 0 | 0 | 0 | 0
  Blue | 7 | 2 | 5 | 14
  Brown | 6 | 13 | 6 | 25
  Hazel | 3 | 1 | 4 | 8
  Green | 1 | 1 | 2 | 4
  Gray | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of ADX-102 on Ocular Discomfort Using the Ora Calibra® Ocular Discomfort Scale.
Description: Change from baseline of ADX-102 on ocular discomfort in subjects with dry eye disease using the Ora Calibra® Ocular Discomfort Scale (0 = least, 4 = most), where a higher score is indicative of a worse outcome. The intervention was administered bilaterally.
Time Frame: Efficacy assessment period (Day 1 through Day 29), Day 29 reported.
Population: Intent-to-treat population with observed data only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADX-102 Ophthalmic Solution (0.1%) | ADX-102 Ophthalmic Solution (0.5%) | ADX-102 Ophthalmic Lipid Solution (0.5%)
Number analyzed (Participants) | 16 | 12 | 11
units on a scale | -0.81 (0.98) | -0.75 (0.75) | -0.82 (1.33)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately four weeks.
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | ADX-102 Ophthalmic Solution (0.1%) | ADX-102 Ophthalmic Lipid Solution (0.5%)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 17/17 | 8/17 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-102 Ophthalmic Solution (0.5%) (N=17) | ADX-102 Ophthalmic Solution (0.1%) (N=17) | ADX-102 Ophthalmic Lipid Solution (0.5%) (N=17)
Instillation site irritation (General disorders) | 17 (17) | 8 (8) | 16 (16) — Transient and self-limiting instillation site irritation that resolved in all cases.
Instillation site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03162783/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT03162783/SAP_003.pdf